CLINICAL TRIAL: NCT01011933
Title: A Phase II Evaluation of AZD6244 (NSC #748727) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Selumetinib in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01958; NCI-2011-01958 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0229H; CDR0000651456; GOG-0229H (Other: NRG Oncology); GOG-0229H (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Blood and archived tumor tissue samples are collected for biomarker studies.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase II trial is studying how well selumetinib works in treating patients with recurrent or persistent endometrial cancer that has come back or is persistent. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of AZD6244 (selumetinib) for patients with recurrent or persistent endometrial cancer with the frequency of patients who survive progression-free for at least 6 months after initiating therapy or have objective tumor response.

II. To determine the nature and degree of toxicity of AZD6244 as assessed by CTCAE v3.0 in this cohort of patients.

SECONDARY OBJECTIVE:

I. To determine the duration of progression-free survival and overall survival.

EXPLORATORY OBJECTIVES:

I. To explore the associations between select biomarkers and response to AZD6244 (progression-free survival status >6 months and objective tumor response), measures of clinical outcome (progression-free survival and overall survival) or disease status including histologic cell type.

II. Mutations and single nucleotide polymorphisms in BRAF, KRAS2, FGFR2, PI3KCA, AKT1, AKT2, AKT3 and PTEN in DNA from formalin-fixed and paraffin-embedded (FFPE) tumor and/or normal blood cells.

III. Immunohistochemical expression of ERK, pERK, GSK3betta, pGSK3betta, PR-A, PR-B, pPR, ER-alpha, ER-beta, BRAF, KRAS, PTEN, EGFR, pEGFR, EGF, PELP1 and MTA1s in FFPE tumor.

IV. To explore the relationship among the panel of biomarkers evaluated in this cohort including mutations and single nucleotide polymorphisms in BRAF, KRAS2, FGFR2, PI3KCA, AKT1, AKT2, AKT3 and PTEN as well as immunohistochemical expression of ERK, pERK, GSK3betta, pGSK3betta, PR-A, PR-B, pPR, ER-alpha, ER-beta, BRAF, KRAS, PTEN, EGFR, pEGFR, EGF, PELP1 and MTA1s.

OUTLINE: This is a multicenter study.

Patients receive selumetinib orally (PO) twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Blood and archived tumor tissue samples are collected for biomarker studies.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed* endometrial epithelial carcinoma, including any of the following cell types:

  * Endometrioid adenocarcinoma
  * Serous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Adenocarcinoma not otherwise specified
  * Mucinous adenocarcinoma
  * Squamous cell carcinoma
  * Transitional cell carcinoma
  * Mesonephric carcinoma
* Recurrent or persistent disease that is refractory to curative therapy or established treatments
* Measurable disease, defined as ≥ 1 lesion that can be measured in ≥ 1 dimension (longest dimension to be recorded)

  * Each lesion must be ≥ 20 mm when measured by conventional techniques (palpation, plain x-ray, CT scan, or MRI) OR ≥ 10 mm when measured by spiral CT scan
* Must have ≥ 1 target lesion to be used to assess response, as defined by RECIST criteria

  * Tumors within a previously irradiated field are designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days following completion of radiotherapy
* Must have received 1 prior chemotherapeutic regimen for the management of endometrial carcinoma

  * Chemotherapy administered as a radiosensitizer in conjunction with primary radiotherapy is considered a systemic chemotherapy regimen
* Not eligible for a higher priority GOG protocol, if one exists (e.g., any active phase III GOG protocol for the same patient population)
* No prior or concurrent CNS disease (treated or untreated) by physical examination, including primary brain tumor or brain metastases
* GOG performance status (PS) 0-2 (for patients who received 1 prior treatment regimen)
* GOG PS 0-1 (for patients who received 2 prior treatment regimens)
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* PT/INR ≤ 1.5 OR in-range INR (between 2 and 3) if patient is on a stable dose of therapeutic warfarin
* PTT ≤ 1.5 times ULN
* Oxygen saturation ≥ 88% on room air
* QTc < 450 msec by EKG
* LVEF normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* No neuropathy (sensory or motor) > grade 1
* No active infection requiring antibiotics

  * Uncomplicated urinary tract infection allowed
* No other invasive malignancy within the past 5 years except for nonmelanoma skin cancer
* No serious, non-healing wound, ulcer, or bone fracture
* No history of abdominal fistula or gastrointestinal perforation
* No intra-abdominal abscess within the past 28 days
* No active bleeding or pathological condition that would carry a high risk of bleeding (e.g., bleeding disorder, coagulopathy, or tumor involving major vessels)
* No seizures not controlled with standard medical therapy
* No clinically significant cardiovascular disease including, but not limited to, any of the following:

  * Uncontrolled hypertension, defined as systolic BP > 140 mm Hg or diastolic BP > 90 mm Hg
  * Myocardial infarction or unstable angina within the past 6 months
  * NYHA class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication, including atrial fibrillation requiring rate-controlling medication
  * Peripheral vascular disease ≥ grade 2
  * Cerebrovascular accident (i.e., CVA, stroke), transient ischemic attack, or subarachnoidal hemorrhage within the past 6 months
* No evidence of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row) by EKG
* Concurrent low molecular weight heparin for treatment of venous thromboembolic disease allowed provided patient is considered clinically stable on this regimen
* Recovered from prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* At least 3 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 3 weeks since other prior therapy directed at the malignant tumor, including immunologic agents
* One prior cytotoxic regimen for the management of recurrent or persistent endometrial disease allowed
* No prior non-cytotoxic chemotherapy for the management of endometrial cancer, except hormonal therapy
* No prior anticancer therapy that contraindicates study therapy
* No prior MEK inhibitor AZD6244 or other specific MEK/ERK/MAPK pathway targeted therapy
* No prior chemotherapy for any abdominal or pelvic tumor other than for the treatment for endometrial cancer within the past 5 years

  * Prior adjuvant chemotherapy for localized breast cancer allowed provided it was completed > 3 years ago AND the patient remains free of recurrent or metastatic disease
* No prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of endometrial cancer within the past 5 years

  * Prior radiotherapy for localized cancer of the breast, head and neck, or skin is allowed provided it was completed > 3 years ago AND the patient remains free of recurrent or metastatic disease
* No concurrent medication that may prolong the QTc interval
* No other concurrent investigational therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — NRG Oncology
Locations (72):
- United States (72):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Coleman RL, Sill MW, Thaker PH, Bender DP, Street D, McGuire WP, Johnston CM, Rotmensch J. A phase II evaluation of selumetinib (AZD6244, ARRY-142886), a selective MEK-1/2 inhibitor in the treatment of recurrent or persistent endometrial cancer: an NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2015 Jul;138(1):30-5. doi: 10.1016/j.ygyno.2015.04.005. Epub 2015 Apr 14. PMID 25887099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study initially opened 9/8/2009 and enrolled 28 participants. It was suspended on 5/17/2010 and re-opened 5/2/2011, enrolling an additional 26 participants until it was closed on 10/24/2011.
Period: Overall Study
Arm/Group | Treatment (Selumetinib)
Started | 54 (total enrolled)
Completed | 50 (total eligible and evaluable)
Not Completed | 4
Not completed — Wrong cell type | 1
Not completed — Improper pre-protocol Rx | 1
Not completed — Inadequate pathology | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: total number of eligible and evaluable participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.7)
Age, Customized [Number; unit: participants]
  40-49 years | 4
  50-59 years | 15
  60-69 years | 18
  70-79 years | 11
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 50
Cell Type [Number; unit: participants]
  Clear cell carcinoma | 1
  Endometrioid adenocarcinoma | 31
  Mixed epithelial carcinoma | 10
  Serous adenocarcinoma | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With or Without Progression-free Survival for > 6 Months by Response Evaluation Criteria for Solid Tumors (RECIST)
Description: Number of participants who survived progression-free for more than 6 months.
  Progression is defined using Response Evaluation Criteria for Solid Tumors (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions in the opinion of the treating physician, or global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression.
Time Frame: > 6 months from study entry
Measure: Number; unit: participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 50
participants
  without progression-free survival | 39
  with progression-free survival | 11

2. Primary Outcome: Objective Tumor Response Rate Assessed by RECIST
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST) Criteria: Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Normalization of CA125, if elevated at study entry, is required; Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD; Increasing Disease is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry; Stable Disease is any condition not meeting the above criteria.
Time Frame: From study entry, assessed up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 50
participants
  Complete Response | 1
  Increase Disease | 23
  Partial Response | 2
  Stable Disease | 13
  Indeterminate | 11

3. Primary Outcome: Participants With Severity of Adverse Effects as Assessed by CTCAE v3.0
Time Frame: Each cycle during treatment and 30 days after the last treatment.
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52
Participants
  Leukopenia | 39 | 11 | 2 | 0 | 0 | 0
  Thrombocytopenia | 48 | 4 | 0 | 0 | 0 | 0
  Neutropenia | 45 | 3 | 2 | 2 | 0 | 0
  Anemia | 21 | 10 | 16 | 4 | 1 | 0
  Auditory/Ear | 51 | 0 | 1 | 0 | 0 | 0
  Cardiac | 45 | 2 | 2 | 3 | 0 | 0
  Coagulation | 51 | 0 | 0 | 1 | 0 | 0
  Constitutional | 16 | 18 | 10 | 8 | 0 | 0
  Dermatologic | 16 | 13 | 18 | 5 | 0 | 0
  Gastrointestinal | 9 | 18 | 19 | 6 | 0 | 0
  Genitourinary/Renal | 50 | 0 | 1 | 1 | 0 | 0
  Hemorrhage | 47 | 4 | 0 | 0 | 0 | 1
  Hepatobiliary | 51 | 0 | 0 | 0 | 0 | 1
  Infection | 51 | 0 | 0 | 0 | 1 | 0
  Lymphatics | 31 | 10 | 7 | 4 | 0 | 0
  Metabolic | 34 | 9 | 3 | 6 | 0 | 0
  Neuropathy | 49 | 2 | 0 | 1 | 0 | 0
  Other Neurological | 44 | 5 | 0 | 3 | 0 | 0
  Ocular/Visual | 48 | 1 | 2 | 1 | 0 | 0
  Pain | 33 | 8 | 6 | 5 | 0 | 0
  Pulmonary | 40 | 6 | 3 | 3 | 0 | 0
  Sexual/Reproductive | 51 | 0 | 2 | 0 | 0 | 0
  Vascular | 51 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Duration of Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle for the first 6 months; then every 3 months thereafter for up to 5 years
Population: Eligible and treated patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 52
months | 2.3 [1.7 to 5.6]

5. Secondary Outcome: Duration of Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 52
months | 8.5 [3.5 to 15.5]

6. Other Pre Specified Outcome: Number of Participants Off Study Therapy for Each Reason Specified.
Time Frame: from study entry until end of study treatment, up to 5 years.
Measure: Number; unit: participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 50
participants
  Disease progression | 32
  Refused further treatment | 5
  Toxicity as permitted | 6
  Death | 2
  Unspecified | 2
  Other - MD decision | 1
  Other - AZD6244 contraindicated w/Amiodarone | 1
  Other - PT never received any study drug | 1

7. Other Pre Specified Outcome: Patient Vital Status
Description: Patients alive or dead after 24 months from time of study entry.
Time Frame: Study entry up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 50
participants
  Alive, without disease progression | 7
  Alive, with disease progression | 4
  Dead, from disease | 37
  Dead, from undetermined cause | 1
  Dead, unspecified | 1

ADVERSE EVENTS:
Time Frame: Adverse Events(AEs) are reported up to 30 days after last treatment. Late AEs can be reported up to 5 years after patient enrollment.
Arm/Group | Treatment (Selumetinib)
Serious Adverse Events (participants affected / at risk) | 32/50
Other Adverse Events (participants affected / at risk) | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=50)
Leukocytes (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 3
Death No Ctcae Term - Death Nos (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Liver Dysfunction (Hepatobiliary disorders) | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 1
Ocular/Visual - Other (Eye disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Vaginitis (Reproductive system and breast disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=50)
Neutrophils (Blood and lymphatic system disorders) | 8
Platelets (Blood and lymphatic system disorders) | 7
Leukocytes (Blood and lymphatic system disorders) | 13
Hemoglobin (Blood and lymphatic system disorders) | 35
Hypotension (Cardiac disorders) | 3
Ptt (Vascular disorders) | 3
Weight Gain (General disorders) | 5
Fever (General disorders) | 7
Rigors/Chills (General disorders) | 3
Fatigue (General disorders) | 38
Insomnia (General disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 15
Rash (Skin and subcutaneous tissue disorders) | 24
Dry Skin (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Heartburn (Gastrointestinal disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 4
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 21
Anorexia (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 34
Diarrhea (Gastrointestinal disorders) | 29
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 3
Edema: Limb (Blood and lymphatic system disorders) | 23
Edema: Head And Neck (Blood and lymphatic system disorders) | 6
Ast (Metabolism and nutrition disorders) | 10
Creatinine (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Alt (Metabolism and nutrition disorders) | 7
Alkaline Phosphatase (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Mood Alteration - Depression (Nervous system disorders) | 6
Mood Alteration - Anxiety (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Neuropathy-Sensory (Nervous system disorders) | 8
Blurred Vision (Eye disorders) | 5
Pain: Extremity-Limb (General disorders) | 6
Pain: Back (General disorders) | 8
Pain: Joint (General disorders) | 6
Pain: Abdominal Pain Nos (General disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less